CLINICAL TRIAL: NCT02166190
Title: Randomized Controlled Trial Comparing Radiofrequency Ablation and Stenting vs. Stenting Alone for Biliary Obstruction Due to Unresectable Cholangiocarcinoma and Pancreatic Cancer
Brief Title: RFA RCT for Pancreatic or Bile Duct Cancer
Acronym: RFARCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment was feasibly not going to be reached.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1403014843
Record Dates: First submitted 2014-06-11; First posted 2014-06-18 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Unresectable Pancreatic Cancer; Cholangiocarcinoma Non-resectable
Keywords: Pancreatic cancer; cholangiocarcinoma; radiofrequency ablation
MeSH Terms: conditions — Pancreatic Neoplasms; Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency Ablation (EndoHbp probe) (Experimental): Radiofrequency Ablation using EndoHPB Probe
  Interventions: Procedure: Radiofrequency Ablation using EndoHPB Probe
- Stenting only (Active Comparator): Stenting only
  Interventions: Procedure: Stenting only

INTERVENTIONS:
Procedure: Radiofrequency Ablation using EndoHPB Probe — Radiofrequency Ablation using EndoHPB Probe
  Arms: Radiofrequency Ablation (EndoHbp probe)
Procedure: Stenting only — Stenting only
  Arms: Stenting only

SUMMARY:
Malignant obstructive jaundice is a common complication of advanced stage pancreatic adenocarcinoma and cholangiocarcinoma. Over 50% of common bile duct (CBD) obstructions are due to malignancy, and the majority of neoplasms are unresectable at the time of diagnosis. Biliary drainage with placement of self-expanding metal stents (SEMSs) for palliation is the therapy of choice in this set of patients. Conventional stent placement provides palliation for a limited duration only and these subjects come back with obstructive jaundice. Due to age, comorbidities, malignant disease status, it is better to conduct reduced number of therapeutic endoscopies to reduce the number of complications. Additionally, only biliary stenting itself may provide only palliation, and not increase the duration of survival.

Currently, there are only two therapies. Recently, photodynamic therapy (PDT) has been evaluated as a palliative and potential neoadjuvant modality. Therefore if RFA confers similar benefits, then it may potentially be used as an alternative to PDT, given the lower adverse event profile. More recently, RFA has been recognized for its potential in palliative treatment of malignant biliary strictures. Based on the published data, RFA provides palliation and seems to increase survival duration in pancreatic cancer. Our own limited experience shows the same. The goal of this randomized controlled trial is to definitely confirm the benefit of Radiofrequency ablation (RFA) in providing increased survival time and quality of life in patients with non-resectable cholangiocarcinoma and pancreatic cancer. These benefits will improve clinical practice by making RFA the new standard of care for unresectable cholangiocarcinoma (CCA) and pancreatic cancer (PC). It will also enhance scientific knowledge by opening the door for new opportunities, e.g. RFA as a potential use for neoadjuvant therapy or as a downstaging agent for surgically resectable patients.

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PC) is a deadly disease. It remains the fourth most common cause of death from cancer in the USA and one of the deadliest cancers in the world. Although treatments have improved, average PC 5-year survival is around 5%. Malignant obstructive jaundice is a common complication of advanced stage pancreatic adenocarcinoma. Over 50% of common bile duct (CBD) obstructions are due to malignancy, and the majority of neoplasms are unresectable at the time of diagnosis.

Biliary drainage with placement of self-expanding metal stents (SEMS) for palliation is the therapy of choice in this set of patients. Metal stenting results in biliary decompression in greater than 80% of cases with a lower complication rate than surgery. When compared to plastic stents, SEMSs present a significantly reduced risk of recurrent biliary obstruction. SEMSs are also more cost effective than plastic stents in patients with a life expectancy of longer than 4 months. Despite their numerous benefits, SEMS become occluded in up to 50% of patients in the first 6-8 months. Covered SEMSs are not resistant to tumor overgrowth or sludge formation and thus stent occlusion results in increased morbidity and mortality.

This relief is temporary since stents tend to become obstructed. More recently, RFA has been recognized for its potential in palliative treatment of malignant biliary strictures.

Photodynamic therapy (PDT) has been previously evaluated as a palliative and potential neoadjuvant modality in patients with biliary obstruction from cholangiocarcinoma. Therefore if RFA confers similar benefits, then it may potentially be used as in a similar manner to PDT, in addition given the lower adverse event profile, it may confer a greater patient tolerance. EndoHPB, the intervention arm, is an endoscopic bipolar catheter designed to ablate tissue in malignant tumors within luminal structures, such as the biliary tree or pancreatic ducts. By using radiofrequency (RF) energy to heat the tissue in the duct prior to insertion of the stent, the surrounding tissue becomes coagulated and this may delay tumor growth and the time before the stent lumen becomes blocked. Thereby, allowing increased periods between the need for intervention and further stent deployment. If EndoHPB use of luminal RF is demonstrated to be effective in luminal tumor ablation, it may have an additional role as a form of neoadjuvant therapy in pancreatic cancer. RFA uses a high frequency alternating current to generate heat and achieve coagulative necrosis when in contact with tissue. Within the bile duct, RFA appears to be safe and may result in decreased benign epithelial hyperplasia and tumor ingrowth. Two recent studies have shown efficacy and safety of RFA in advanced pancreatic and cholangiocarcinoma. Subsequently, retrospective collection of data from a cohort of 26 patients treated with endobiliary RFA for malignant biliary obstruction in our Institution confirmed the safety of this approach and suggested a potential survival benefit at 90 and 180 days post treatment compared to matched controls.

A pilot study was initiated and IRB approved at the Weill Cornell Medical College in 2011 with primary investigator Dr. Michel Kahaleh. The study was closed in Nov 2013 as the results showed that RFA significantly increased the bile duct diameter. Analysis also showed that survival duration was slightly increased in the Pancreatic Cancer group.

* Hypothesis: Luminal application of RF energy using EndoHPB in the bile duct of patients with cholangiocarcinoma or pancreatic cancer provides ablation of tumor causing biliary obstruction(s). Effectiveness will assessed by looking at the change in diameter(s), on cholangiography and assess time till stent occlusion.
* Study Design: Randomized, Controlled, 2- arm, Non-Blinded, Randomised controlled trial Treatment group: Endoscopic retrograde cholangiopancreatography (ERCP) with RFA and biliary stenting.

Control group: ERCP with biliary stenting only

* Primary outcome measure: is survival time, measured from the date of randomization until the date of death or the last date the patient was known to be alive.
* Secondary outcome measure: Number of Participants with Adverse Events. To assess safety of an endoscopic bipolar radiofrequency catheter (EndoHPB) in the management of unresectable cholangiocarcinoma and pancreatic cancer.
* Condition : - Unresectable Cholangiocarcinoma or Pancreatic Cancer
* Intervention: Endoscopic radiofrequency ablation using the ENDOHPB probe.

ELIGIBILITY:
Inclusion Criteria:

- Either gender greater than or equal to 18 years of age.

* Pancreatic cancer or cholangiocarcinoma unsuitable for surgical resection. Criteria of unresectability being based on 1) metastatic disease or 2) locally advanced. Subjects that are deemed to be unresectable will be determined by a surgeon or treating oncologist.
* Biliary obstruction
* Subjects capable of giving informed consent
* Life expectancy of at least 6 months

Exclusion Criteria:

- Exclusion Criteria

* Cardiac Pacemaker
* Patient unstable for ERCP or has failed ERCP (endoscopic retrograde cholangiopancreatography )
* Inability to give informed consent
* Uncorrected coagulopathy
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-06; Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
Clinical Success- composite | 1 year
  Clinical Success Composite of Stent patency, serum bilirubin and general quality of life measured at 3 months, 6 months, 9 months and 12 months as well as survival duration.

SECONDARY OUTCOMES:
Mutational Profile of DNA post interventional procedure | 1 year
  Mutational profile of DNA using FISH (Fluorescence in situ hybridization) analysis on brushings of bile duct after RFA procedure to further understand the implications at the cellular and genetic level at 1 month, 3 months, 6 months, and 9 months

OTHER OUTCOMES:
Safety Profile and Quality of Life | 1 year
  Number of adverse events, severity and frequency of adverse events and relatedness to procedure within 30 days of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Reem Z Sharaiha, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No IPD sharing